CLINICAL TRIAL: NCT04829799
Title: Effect of Intracameral Phenylephrine/Ketorolac on Intraoperative Pain
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Per study team, the study will not proceed
Sponsor: University of Florida (Other)
Collaborators: Omeros Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB202002831 -A; OCR40493 (Other: UF OnCore)
Record Dates: First submitted 2021-03-31; First posted 2021-04-02 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Pain Reduction
MeSH Terms: interventions — Phenylephrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control Group (Active Comparator): Subjects will receive intracameral 1% preservative-free lidocaine following paracentesis
  Interventions: Drug: 1% preservative-free lidocaine
- Study Experimental Group (Experimental): Subject will receive Omidria (phenylephrine and ketorolac (1.0%/0.3%) added to the ophthalmic irrigating solution during the cataract extraction procedure
  Interventions: Drug: Phenylephrine 1.0%/ Ketorolac 0.3%

INTERVENTIONS:
Drug: 1% preservative-free lidocaine — Instillation of intracameral lidocaine after initial paracentesis incision.
  Arms: Control Group
Drug: Phenylephrine 1.0%/ Ketorolac 0.3% — Instillation of Omidria irrigation solution after paracentesis incision and in irrigation solution.
  Arms: Study Experimental Group

SUMMARY:
To compare the effect of intraoperative intracameral Omidria (Phenylephrine and Ketorolac 1.0%/0.3%) verses 1% Lidocaine on pain reduction during and after cataract surgery.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a cataract in the surgical eye

Exclusion Criteria:

* Patients that have previously exhibited sensitivities to acetylsalicylic acid, phenylacetic acid derivative, and other nonsteroidal anti-inflammatory drugs (NSAIDs)
* Those with a past medical history of asthma
* Those systemically using opioids or nonsteroidal anti-inflammatory drugs
* Those prescribed additional topical mydriatics, topical steroids, pilocarpine, or prostaglandins in the week preceding surgery
* Those with a history of alpha-1-adrenergic antagonist use
* Those with excisional, intraocular surgery in the planned surgical eye in the preceding year
* Those with a history of iris damage
* Those requiring iris expanding device or those with an acute or chronic uncontrolled eye condition, or those unable to effectively remember surgery or complete the post-operative assessment.
* Additionally, individuals less than 21 will be excluded.

Ages: 40 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-02 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale to measure pain | Day 1 of operation
  Measurement of pain intensity by mean visual analog scale (VAS) pain scores from 0 (no pain) to 10 (extreme pain) during operation

CONTACTS AND LOCATIONS:
Overall Officials: Eric Grieser, MD, Principal Investigator — University of Florida

IPD SHARING:
Plan to Share IPD: No